CLINICAL TRIAL: NCT06192264
Title: A Phase III Randomized, Double-blind, Placebo-controlled, Multi-center Study to Evaluate Safety and Efficacy of ASC40 (Denifanstat) Tablets in Subjects With Moderate to Severe Acne Vulgaris
Brief Title: A Study to Evaluate the Safety and Efficacy of ASC40 (Denifanstat) Tablets in the Treatment of Patients With Moderate to Severe Acne Vulgaris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ascletis Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Ascletis Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ASC40-303
Record Dates: First submitted 2023-12-14; First posted 2024-01-05 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-05

CONDITIONS: Acne
Keywords: Acne; ASC40
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ASC40 dose 1 (Experimental): ASC40 dose 1 84 days of treatment
  Interventions: Drug: ASC40
- ASC40 Placebo (Placebo Comparator): ASC40 Placebo 84 days of treatment
  Interventions: Drug: ASC40

INTERVENTIONS:
Drug: ASC40 — ASC 40 tablets orally once daily

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled Phase III study to evaluate the efficacy and safety of ASC40 (Denifanstat) tablets compared to placebo in the treatment of patients with moderate to severe acne vulgaris. The proposed plan for this trial is to enroll subjects who are 18-40 years of age (including borderline values), with a diagnosis of moderate to severe acne vulgaris, and an Investigator's Global Assessment (IGA) graded as moderate (grade 3) or severe (grade 4). 480 subjects were planned to be enrolled in the trial and placebo groups, with all subjects randomly assigned in a 1:1 ratio to receive either ASC40 (denifanstat) tablets dose 1 or placebo, administered orally once daily (taken after dinner) for 12 weeks.

There will be a total of 6 visits for screening and follow-up. The tests required by the program included routine blood tests, blood biochemistry, lipid profile, pregnancy test and urine routine, etc..

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years (inclusive of threshold), gender is not limited.
* Subjects have an Investigator's Global Assessment (IGA) score of 3 or 4 (i.e., moderate or severe).
* Men of childbearing potential and women of childbearing potential willing to use effective contraception from the time of signing the informed consent until 3 months after the last dose of the investigational drug; women of childbearing potential include premenopausal women and women within 2 years of menopause. Women of childbearing potential must have a negative pregnancy test result within ≤ 7 days prior to the first dose of the investigational drug.
* Subjects are willing and able to complete the study, are able to understand and comply with the study requirements, adhere to the study required restrictions and related tutorials, use the investigational drug as prescribed, and are followed up according to the study plan.

Exclusion Criteria:

* Known hypersensitivity to the ingredients of ASC40 (Denifanstat) tablets or to any of the excipients.
* Presence of cystic acne at screening.
* Patients with secondary acne such as occupational acne (e.g., chloracne) and corticosteroid-induced secondary acne (e.g., chloracne or drug-induced acne)
* Patients with other significant coexisting skin conditions that may affect the evaluation of facial acne efficacy or require co-treatment, such as solardermatitis, psoriasis, seborrheic dermatitis, rosacea, folliculitis, eczema, etc..
* Thicker facial hair, which has been assessed by researchers to impede accurate assessment of acne vulgaris grades or lesion counts

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 480 (Actual)
Dates: Start 2024-01-23 (Actual); Primary Completion 2025-05-19 (Actual); Study Completion 2025-05-19 (Actual)

PRIMARY OUTCOMES:
Percentage of treatment success based on investigator's global assessment (IGA) in each group of subjects | At Week 12 of treatment.
  Percentage of treatment success subjects in each group based on investigator's global assessment (IGA) at Week 12 (treatment success defined as an IGA grade of 0 or 1, and a ≥2-grade decrease in IGA grade from baseline)
Percentage change in total skin lesion counts compared to baseline ineach group of subjects | At Week 12 of treatment.
  Percentage change in total skin lesion counts compared to baseline for subjects in each group at Week 12
Percentage change in the count of inflammatory skin lesions compared to baseline in each group of subjects | At Week 12 of treatment.
  Percentage change in inflammatory skin lesion counts compared to baseline for subjects in each group at Week 12

SECONDARY OUTCOMES:
Percentage change in non-inflammatory lesion counts compared to baseline for each group of subjects | At Week 12 of treatment.
  Percentage change in non-inflammatory lesion counts compared to baseline for subjects in each group at Week 12
Absolute change in total skin lesion counts compared to baseline for each group of subjects | At Week 12 of treatment.
  Absolute change in total skin lesion counts compared to baseline for each group of subjects at Week 12
Absolute change in inflammatory skin lesion counts compared to baseline in each group of subjects | At Week 12 of treatment.
  Absolute change in inflammatory skin lesion counts compared to baseline in each group of subjects at Week 12

CONTACTS AND LOCATIONS:
Locations (41):
- China (41):
  - The First Affiliated Hospital of Bengbu Medical University, Bengbu, Anhui
  - The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - The First Affiliated Hospital of Wannan Medical College, Wuhu, Anhui
  - The Second Affiliated Hospital of Wannan Medical College, Wuhu, Anhui
  - Beijing Tsinghua Changgeng Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Dermatology Hospital of Southern Medical University, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The Fifth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Shenzhen Hospital, The University of Hong Kong, Shenzhen, Guangdong
  - The Affiliated Hospital of Guangdong Medical University, Zhanjiang, Guangdong
  - Guilin Medical College Affiliated Hospital, Guilin, Guangxi
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangzhou
  - Shenzhen People's Hospital, Shenzhen, Guangzhou
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Nanyang First People's Hospital, Nanyang, Henan
  - Tongji Hospital Affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Wuhan Central Hospital, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Changzhou First People's Hospital, Changzhou, Jiangsu
  - Lianyungang First People's Hospital, Lianyungang, Jiangsu
  - The First Affiliated Hospital of Gannan Medical College, Ganzhou, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Huashan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Skin Disease Hospital, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Xi'an Medical College, Xi’an, Shanxi
  - The Second Affiliated Hospital of Xi'an Jiaotong University School of Medicine, Xi’an, Shanxi
  - Chengdu Second People's Hospital, Chengdu, Sichuan
  - Suining Central Hospital, Suining, Sichuan
  - Tianjin Medical University General Hospital, Tianjing, Tianjing
  - Hangzhou First People's Hospital, Hangzhou, Zhejiang
  - Hangzhou Third People's Hospital, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital Affiliated to Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Ningbo Second Hospital, Ningbo, Zhejiang
  - The First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - The Fourth Affiliated Hospital of Zhejiang University School of Medicine, Yiwu, Zhejiang

IPD SHARING:
Plan to Share IPD: No